CLINICAL TRIAL: NCT04679350
Title: A Multi Center, Randomized, Double-blind, Parallel Design, Phase 2 Study to Evaluate the Efficacy and Safety of hzVSFv13 Compared to Standard of Care After Intravenous(IV) Administration With Add-on Standard of Care in COVID-19 Moderate to Severe Patients
Brief Title: Efficacy and Safety of hzVSFv13 in Patients With COVID-19 Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A new study combining Phase III clinical trials has been planned.
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM_hzVSF_v13-0004
Record Dates: First submitted 2020-12-21; First posted 2020-12-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard of care + 3 doses of hzVSF-v13 50 mg/dose IV (Experimental): Standard of care + 3 doses of hzVSF-v13 50 mg/dose IV
  Interventions: Drug: hzVSF-v13
- Standard of care + 3 doses of hzVSF-v13 200 mg/dose IV (Experimental): Standard of care + 3 doses of hzVSF-v13 200 mg/dose IV
  Interventions: Drug: hzVSF-v13
- Standard of care + 1 dose of hzVSF-v13 200 mg/dose IV + 2 doses of the placebo (Experimental): Standard of care + 1 dose of hzVSF-v13 200 mg/dose IV + 2 doses of the placebo
  Interventions: Drug: hzVSF-v13
- Standard of care + 3 doses of the placebo to match hzVSF-v13 (normal saline) (Placebo Comparator): Standard of care + 3 doses of the placebo to match hzVSF-v13 (normal saline)
  Interventions: Drug: Placebo (Normal saline solution)

INTERVENTIONS:
Drug: hzVSF-v13 — Drug: hzVSF-v13 Dosage form: hzVSF-v13 40mg/mL in a 5mL vial Frequency: Dose at Day 1, 3, 7 Other names: a humanized monoclonal antibody (mAb)
  Other Names: a humanized monoclonal antibody (mAb)
  Arms: Standard of care + 1 dose of hzVSF-v13 200 mg/dose IV + 2 doses of the placebo; Standard of care + 3 doses of hzVSF-v13 200 mg/dose IV; Standard of care + 3 doses of hzVSF-v13 50 mg/dose IV
Drug: Placebo (Normal saline solution) — Dosage form: 0.9% NaCl solution Frequency: Dose at Day 1, 3, 7
  Other Names: 0.9% Normal saline
  Arms: Standard of care + 3 doses of the placebo to match hzVSF-v13 (normal saline)

SUMMARY:
To explore the efficacy and confirm the safety of the concomitant administration of the standard of care and hzVSF-v13 in patients with COVID-19 infection

DETAILED DESCRIPTION:
A Multi center, Randomized, Double-blind, Parallel design

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged at least 19 years at screening
2. Those who have been admitted or scheduled to be admitted due to a diagnosis with COVID-19 by RT-PCR test within 4 days prior to screening
3. Patients whose findings of COVID-19 pneumonia have been confirmed by radiographic tests (CT and X-ray) at screening (e.g., ground glass opacity (GGO), crazy-paving pattern, or consolidation)
4. Those who fall under the following at screening:

   - Patients identified as moderate: Oxygen saturation in the atmosphere (SpO2) >93% (to be confirmed with respiratory rate ≥20/min or pulse rate ≥90 beats/min secondarily)
   * Patients identified as severe: Oxygen saturation in the atmosphere (SpO2) ≤93% or PaO2/FiO2 <300 (respiratory rate ≥30/min or pulse rate ≥125 beats/min secondarily)
5. Those who have voluntarily provided a written consent to participate in this clinical study

Exclusion Criteria:

1. Individuals with a clinically significant history of hypersensitivity reactions to the components of hzVSF-v13, drugs containing components of the same class, or other drugs (aspirin, non-steroidal anti-inflammatory drugs, antibiotics, etc.)
2. Individuals with a severe at screening

   - Breathing disorder that requires treatment of one or more of the following: Oxygen therapy using high-flow nasal cannula (HFNC), Noninvasive positive pressure ventilation (NIV), invasive mechanical ventilation, ECMO, Clinical diagnosis of respiratory failure

   - Shock (Systolic <90mmHg or diastolic <60mmHg, or in case need a blood pressure booster)

   - Multiple organ failure
3. Patients with pneumonia other than due to the novel coronavirus (SARS-CoV-2) infection (e.g., influenza virus pneumonia, bacterial pneumonia, and fungal pneumonia)
4. Patients with severe heart failure (NYHA Class III or higher)
5. Pregnant women
6. Men or women of childbearing potential who are planning to become pregnant or do not agree to use one or more of the clinically appropriate methods of contraception below from the first day until 120 days after the last day of investigational product administration

   ① Surgical infertility (e.g., bilateral tubal ligation, vasectomy)

   ② Hormonal contraceptives (Hormone releasing IUD, implantable form, patch, oral hormone)

   ③ Double-barrier method (concomitant use of two of the following: IUD, male or female condom, contraceptive diaphragm, contraceptive sponge, cervical cap, spermicide) Periodic abstinence (e.g., calendar, ovulation date, basal body temperature, post-ovulation methods) and coitus interruptus are not permitted as appropriate contraceptive methods, and effective contraceptive methods must be kept being used during the course of the clinical study.
7. Those who are scheduled to have organ transplantation
8. Those who have laboratory test results that fall under the following values at screening ① ALT or AST ≥5 times the upper limit of normal (ULN)

   ② eGFR < 30 mL/min/1.73m2

   ③ platelets < 50,000/mm3
9. Those who have a positive result for serology (hepatitis B, human immunodeficiency virus [HIV], and hepatitis C tests) at screening
10. Those who administered other investigational products within 30 days prior to the screening visit
11. Others who have been determined to be ineligible to participate in the clinical study according to the investigator's medical opinion

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in the clinical improvement score on an 8-point scale at Day 21 | Day 21
  Descriptive statistics for the changes from baseline in the clinical improvement score on an 8-point scale at Day 21 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon rank-sum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.

SECONDARY OUTCOMES:
Changes from baseline in the clinical improvement score on an 8-point scale at Day 7, Day 14, and Day 28 | Day 7, Day 14, Day 28
  Descriptive statistics for the changes from baseline in the clinical improvement score on an 8-point scale at Day 7, Day 14, and Day 28 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon ranksum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.
Time to discontinuation of oxygen therapy after investigational product administration | Day 28
  The Kaplan-Meier curves for the time to discontinuation of oxygen therapy after investigational product administration shall be presented, and the median time and 95% confidence interval will be presented by treatment group. In addition, a log-rank test shall be performed, if necessary, to test differences of each study group compared to the control group.
Time to recovery* after investigational product administration (days) | Day 28
  *0 to 3 points in the clinical improvement score on an 8-point scale The Kaplan-Meier curves for the time to recovery after investigational product administration shall be presented, and the median time and 95% confidence interval will be presented by treatment group. In addition, a log-rank test shall be performed, if necessary, to test differences of each study group compared to the control group.
Changes from baseline in PaO2/FiO2 at Day 7, Day 14, Day 21, and Day 28 | Day 7, Day 14, Day 21, Day 28
  Descriptive statistics for the changes from baseline in PaO2/FiO2 at Day 7, Day 14, Day 21, and Day 28 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon rank-sum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.
Changes from baseline in the NEWS 2 score at Day 7, Day 14, Day 21, and Day 28 | Day 7, Day 14, Day 21, Day 28
  Descriptive statistics for the changes from baseline in the NEWS 2 score at Day 7, Day 14, Day 21, and Day 28 shall be presented for each treatment group, and a two-sample t-test or the Wilcoxon rank-sum test shall be performed depending on whether the normality assumption is satisfied in order to test differences of each study group compared to the control group.
Mortality at Day 28 and Day 60 after investigational product administration | Day 28, Day 60
  The frequency and percentage for the proportion of subjects who died at Day 28 and Day 60 after investigational product administration shall be presented for each treatment group, and the Pearson's chi-squared test or the Fisher's exact test shall be performed to test differences of each study group compared to the control group.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Yeungnam University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon

IPD SHARING:
Plan to Share IPD: No